CLINICAL TRIAL: NCT02773251
Title: Hyaluronic Acid-Carboxymethylcellulose Reduced Postoperative Bowel Adhesions Following Laparoscopic Urologic Pelvic Surgery: a Prospective, Randomized, Controlled, Single-Blind Study
Brief Title: The Effect of Guardix-solution for the Prevention of Postoperative Intestinal Adhesion and Intestinal Obstruction After Laparoscopic Pelvic Cavity Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bucheon St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Koh Jun Sung, Professor, Bucheon St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XC11DIMI10098H
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer; Postoperative Adhesion
Keywords: Postoperative adhesion; Laparoscopy; Adhesion barrier
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hyaluronic acid-carboxymethylcellulose treatment group (Experimental): the HA/CMC treatment group after laparoscopic pelvic surgery
  Interventions: Drug: hyaluronic acid-carboxymethylcellulose
- control group (No Intervention): the HA/CMC non-treatment group after laparoscopic pelvic surgery

INTERVENTIONS:
Drug: hyaluronic acid-carboxymethylcellulose
  Arms: hyaluronic acid-carboxymethylcellulose treatment group

SUMMARY:
To assess the anti-adhesive effect of treatment with hyaluronic acid-carboxymethylcellulose following laparoscopic pelvic surgery (radical prostatectomy).

DETAILED DESCRIPTION:
Methods This was a prospective, randomized, controlled, single-blind, parallel-group study using HA/CMC (marketed as Guardix-sol®, Hanmi Medicare, Seoul, Korea) in patients who underwent laparoscopic radical prostatectomy between November 2011 and June 2014. All the patients were informed in detail about the aims and the procedures of the study and they signed a written informed consent prior inclusion into the study. The protocol and the written informed consent were approved by the local ethical committee (Catholic Medical Center, Clinical Research Coordinator Center; approval number XC11DIMI10098H).

Subjects Men who were 50-75 years old and diagnosed with prostate cancer were eligible if they were scheduled to undergo laparoscopic radical prostatectomy. Exclusion criteria included any history of abdominal or pelvic surgery, hypersensitivity or an allergic reaction to the study material, pelvic lymph node dissection at the same time as prostatectomy, the presence of surgical site infection or contamination, a history of a medical disease causing bowel adhesion, or a history of severe drug allergies.

Study design and protocol The laparoscopic radical prostatectomy was performed in same surgical procedures and steps by two surgeons (USH and JSK) who have experienced over 150 cases of laparoscopic radical prostatectomy. The laparoscopic radical prostatectomy was performed using the five-port fan-shaped transperitoneal approach. After the introducing the peritoneal cavity, incising the parietal peritoneum between the medial umbilical ligaments are incised and dissection is carried through the fatty alveolar tissue to develop the space of Retzius. After that, the surgical steps are following order (1) incision of the endopelvic fascia; (2) ligation of the dorsal vein complex; (3) division of the bladder neck; (4) dissection of the seminal vesicles; (5) incision of the Denonvillier fascia and control of the lateral pedicles with antegrade neurovascular bundle dissection; (8) apical dissection and division of the dorsal vein and the urethra; (9) urethrovesical anastomosis.

Considering about 30% of dropout rate (under the assumption of 40% difference between HA/CMC treatment group and the control group based on previous similar study, by which the target enrollment for this trial was 60 subjects (30 subjects per group). The sample size was determined assuming a level of significance of α=0.05 (two-side) and a 80% statistical power of test. All patients were randomly assigned to either the HA/CMC treatment group (n=30) or the control group (n=30) using a computer-generated randomization table. The surgeon was blinded to treatment assignments before randomization. Patients were also blinded to their treatment group throughout the study. HA/CMC was applied in all port sites and the peritoneal incision line of the medial umbilical ligament with a single-use applicator attached to a sprayer that allowed for the precise application to the required sites. The amount of HA/CMC applied was 5 ml. Information regarding the duration of illness and medical history were collected at the time of enrollment (V0). Viscera slide ultrasound and plain X-ray were recorded at the time of the operation (V0) and 12 (V1) and 24 week (V2) after the operation.

The primary end point was the difference in excursion distance on viscera slide ultrasound between V0 and V2. The secondary end point was excursion distance on viscera slide ultrasound at V2 and the presence of restriction of viscera slide on ultrasound at V2.

Assessment of efficacy and safety Twelve and 24 weeks after the operation, bowel adhesion to the abdominal wall was evaluated by ultrasound and plain X-rays. We performed viscera slide ultrasound according to a technique that has been previously described. By dividing the abdomen into 5 segments and examining the viscera slide in each segment, a prediction of the extent of the adhesions was made for each patient. At the time of the viscera slide ultrasound, data were also collected on the location of the scars on the abdomen. The main point of interest was the distance of the longitudinal excursion of the selected area in relation to the fixed abdominal wall. Normal viscera sliding movement was defined as equal to or greater than 1 cm of longitudinal movement. Restricted viscera slide was defined as less than 1 cm of longitudinal movement during both normal and exaggerated respiration. The ultrasound was performed by two sonographers who had been well instructed for study assessment. The assessment by ultrasound was double-checked. The sonographer, radiologist and all accessor was blind to the randomization during the all study period.

Statistical Analysis The data for this study are expressed as mean ± standard deviation of the mean. The comparisons of the 2 groups were made using a chi-test, an independent Student's t test, or repeated measure ANOVA. P-values <0.05 were considered significant. Statistical calculations were carried out with IBM SPSS statistics, Version 21 (IBM Corp, Armonk, NY).

ELIGIBILITY:
Inclusion Criteria:

* Men who were 50-75 years old and diagnosed with prostate cancer were eligible if they were scheduled to undergo laparoscopic pelvic surgery (radical prostatectomy).

Exclusion Criteria:

* any history of abdominal or pelvic surgery, hypersensitivity or an allergic reaction to the study material, pelvic lymph node dissection at the same time as prostatectomy, the presence of surgical site infection or contamination, a history of a medical disease causing bowel adhesion, or a history of severe drug allergies.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
the difference in excursion distance on viscera slide ultrasound between V0 and V2. | within the first 6 months after surgery

REFERENCES:
- [Derived] Ha US, Koh JS, Cho KJ, Yoon BI, Lee KW, Hong SH, Lee JY. Hyaluronic acid-carboxymethylcellulose reduced postoperative bowel adhesions following laparoscopic urologic pelvic surgery: a prospective, randomized, controlled, single-blind study. BMC Urol. 2016 Jun 10;16(1):28. doi: 10.1186/s12894-016-0149-3. PMID 27286961